CLINICAL TRIAL: NCT04701619
Title: Immuno-inflammatory Profile and Response to Ischemic Stroke Reperfusion Therapies
Brief Title: Immuno-inflammatory Profile and Response to Ischemic Stroke Reperfusion Therapies (IMMUNOSTROKE)
Acronym: IMMUNOSTROKE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BMR_2020_31
Record Dates: First submitted 2020-11-25; First posted 2021-01-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: All patients undergoing a reperfusion procedure as part of an ischemia stroke will be able to participate in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immuno-inflammatory profile description in patients with ischemic stroke (Other): Patients will be evaluated for inflammatory biomarkers at inclusion, at 24-48 hours of reperfusion treatment , at 72 hours, at 7 days or at discharge if before D7, at discharge if after D7, at 3 months and at 1 year.The biomarkers will be measured using ELISA panels for inflammatory biomarkers
  Interventions: Other: Immuno-inflammatory profile description in patients with ischemic stroke

INTERVENTIONS:
Other: Immuno-inflammatory profile description in patients with ischemic stroke — Patients will be evaluated for inflammatory biomarkers at inclusion, at 24-48 hours of reperfusion treatment , at 72 hours, at 7 days or at discharge if before D7, at discharge if after D7, at 3 months and at 1 year.The biomarkers will be measured using ELISA panels for inflammatory biomarkers

SUMMARY:
IMMUNOSTROKE study aims to describe the immuno-inflammatory and thrombo-inflammatory profiles during the course of AIC management by reperfusion treatment and to monitor changes in these different parameters over time. Post-hoc analyses will make it possible to correlate the immuno-inflammatory and thrombo-inflammatory profiles and their evolution with the clinical outcome in terms of post-AIC functional and cognitive disability.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Presenting with an ACS for which reperfusion therapy is indicated according to European and North American recommendations (IV thrombolysis or mechanical thrombectomy or a combination of both)
* Having received informed information about the study and having signed a consent form to participate in the study (if this is not possible: information and consent from a trusted person or family member if present; emergency inclusion if absent)
* Affiliated with or beneficiary of a social security system

Exclusion Criteria:

* Contraindication to performing a brain MRI (claustrophobia, pacemaker, or other implantable device contraindicating the performance of an MRI)
* Intracranial hemorrhage associated with AIC on initial imaging

Immunosuppressive treatment or corticosteroid therapy at patient admission

* Pre-existing neurological disability limiting neurological assessment at 3 months (mRS>2 at admission)
* Known and diagnosed dementia pre-existing at the time of the AIC
* Absolute or relative contraindication to the injection of gadolinium (history of true allergic reaction or intolerance to gadobutrol, renal failure with creatinine clearance <15mL/min, pregnant or breastfeeding women)
* Patient treated by another institution and referred solely for mechanical thrombectomy
* Patient benefiting from legal protection measures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-09-15 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Immuno-inflammatory profile description in patients with ischemic stroke and eligible for reperfusion treatment | Up to year
  Patients will be evaluated for inflammatory biomarkers at inclusion, at 24-48 hours of reperfusion treatment , at 72 hours, at 7 days or at discharge if before D7, at discharge if after D7, at 3 months and at 1 year.The biomarkers will be measured using ELISA preconfigurated panels for inflammatory biomarkers.